CLINICAL TRIAL: NCT03480321
Title: An Open-Label, Randomized, Three-Treatment, Three-Way Crossover Pharmacokinetic Study of Once Daily PMR Compared to Twice Daily Cilostazol IR Tablets in Healthy Volunteers
Brief Title: Pharmacokinetic Study of Once Daily PMR Compared to Twice Daily Cilostazol IR Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GBL17-001
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Intermittent Claudication
Keywords: Peripheral Artery Disease; Cilostazol; PMR; Extended-Release Tablet of Cilostazol
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — Cilostazol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cilostazol 100 mg (Active Comparator)
  Interventions: Drug: Cilostazol 100 mg
- PMR 150 mg (Experimental)
  Interventions: Drug: PMR 150 mg
- PMR 200 mg (Experimental)
  Interventions: Drug: PMR 200 mg

INTERVENTIONS:
Drug: Cilostazol 100 mg — One immediately-release tablet (Cilostazol 100 mg) at 08:00 and another at 20:00, twice daily oral dose (total daily dose of 200 mg)
  Arms: Cilostazol 100 mg
Drug: PMR 150 mg — Two extended-release tablets (PMR 150 mg) at 08:00, single oral dose (total daily dose of 300 mg)
  Arms: PMR 150 mg
Drug: PMR 200 mg — Two extended-release tablets (PMR 200 mg/tablet) at 08:00, single oral dose (total daily dose of 400 mg)
  Arms: PMR 200 mg

SUMMARY:
The study is designed to evaluate the bioequivalency between the test formulations of extended-release tablet of cilostazol (PMR) administered once-daily and the reference formulation of immediate-release tablet of cilostazol (Cilostazol) administered twice-daily in normal healthy male and female subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 to 45 years of age, inclusive.
* Absence of diseases, such as heart failure, significant kidney impairment or a history of restricted blood flow to the heart, that could affect the study outcomes.
* Having a body mass index (BMI) within normal standard limits (18.5~24.9, inclusive).
* Willing and able to give informed consent to participate in the clinical study and comply with all study procedures, restrictions and attend all visits.

Exclusion Criteria:

* History of bleeding tendency.
* Use of anticoagulant agent(s) within 1 month prior to screening.
* Use of tobacco or nicotine products within 6 months of screening.
* Intake of over the counter or prescription drugs (other than hormonal contraceptives) within 2 weeks prior to randomization.
* On any investigational drug(s) or therapeutic device(s) within 30 days preceding screening; or anticipating use of any of these therapies during the course of the study (other than the study products).
* History of substance abuse, such as alcohol, IV drugs, and inhaled drugs, within 1 year prior to screening.
* Known history of having Acquired Immunodeficiency Syndrome (AIDS) or positive pre-study result of infection with Human Immunodeficiency Virus (HIV); history or positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Pregnant or breast feeding.
* Women of child-bearing potential not using an effective birth control method. Women of child-bearing potential are defined as women physiologically capable of becoming pregnant, UNLESS they meet the following criteria:

  1. Post-menopausal: 12 months of natural (spontaneous) amenorrhea or less than 12 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40IU/L, OR;
  2. 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy, OR;
  3. Using one or more of the following acceptable methods of contraception: surgical sterilization (e.g. bilateral tubal ligation), hormonal contraception (e.g. implantable, injectable, vaginal patch, and oral), and double-barrier methods. Reliable contraception should be maintained throughout the study and for 7 days after study discontinuation.
* Known or suspected hypersensitivity to any ingredient of study drug(s).
* Donated blood or lost more than 150 mL of blood within 3 months prior to randomization or plans to donate blood or plasma within 4 weeks after completion of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve, from time zero to last measureable time point (AUC (0-t)) | 0-72 hours after morning dose
AUC from time zero to infinity (AUC (0-∞)) | 0-72 hours after morning dose

CONTACTS AND LOCATIONS:
Locations (1):
- Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No